CLINICAL TRIAL: NCT05064033
Title: Pragmatic Posterior Capsular Stretch Versus Sleeper Stretch in Subject With Shoulder Pathologies: a Randomized Control Trial (RCT)
Brief Title: Pragmatic Posterior Capsular Stretch Versus Sleeper Stretch in Subject With Shoulder Pathologies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helping Hand Institute of Rehabilitation Sciences (Other)
Responsible Party: Principal Investigator, Keramat Ullah, Principal HHIRS, Helping Hand Institute of Rehabilitation Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Rec.letter/st./2021/20/03/04
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Shoulder Impingement; Shoulder Arthritis; Shoulder Injuries; Shoulder Capsulitis; Shoulder Bursitis; Shoulder Pain Chronic
Keywords: sleeper stretch; shoulder pathologies; Posterior capsular tightness; shoulder range of motion; pragmatic posterior capsular stretch; pragmatic intervention
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Injuries

STUDY DESIGN:
Intervention Model Description: Randomized control trial(double-blind)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): Pragmatic Set of intervention and posterior capsular stretch
  Interventions: Other: Pragmatic Set of intervention and posterior capsular stretch
- GROUP B (Active Comparator): Pragmatic Set of intervention and Sleeper Stretch
  Interventions: Other: Pragmatic Set of intervention and Sleeper Stretch

INTERVENTIONS:
Other: Pragmatic Set of intervention and posterior capsular stretch — Group 1 will receive a pragmatic set of interventions, including Serratus Anterior Stretch,Rotator Cuff Facilitation,Acromilcalavicular joint Mobilization,Stretch of Pectoralis Major and Minor,Thoracic Manipulation and posterior capsular stretch.
  Arms: GROUP A
Other: Pragmatic Set of intervention and Sleeper Stretch — Group 2 will receive a pragmatic set of interventions, including Serratus Anterior Stretch, Rotator Cuff Facilitation, Acromilcalavicular joint Mobilization, Stretch of Pectoralis Major and Minor, Thoracic Manipulation and sleeper stretch.
  Arms: GROUP B

SUMMARY:
The glenohumeral joint is an articulation between the glenoid of the scapula and the head of the humerus that is enclosed by a synovial capsule divided into three main components: anterior, posterior, and the axillary pouch. Symptoms of posterior capsule tightness are linked to altered shoulder biomechanics and impairments which includes glenohumeral internal rotation deficit, incomplete glenohumeral adduction, impaired inferior glenohumeral ligament (IGHL) function, and increased risk of impingement symptoms. In the literature the two techniques available for stretching posterior capsule are pragmatic posterior capsular stretch and sleeper stretch. Pragmatic posterior capsular stretch is therapist administered and sleeper stretch is patient-administered. The work on the pragmatic posterior capsular stretch is more specified and rational to mark the tightness in the posterior capsule.

DETAILED DESCRIPTION:
Shoulder pathologies have been reported as the third most popular musculoskeletal problem after knee and back problems and are relatively common in 1 in 3 individuals in their lifetime and reported shoulder pain once a year. The Popular shoulder complex disorders are tendinopathies, rotator cuff lesions, serratus anterior paralysis, subacromial impingement syndrome, and adhesive capsulitis among these 44-65 percent shoulder disorders, contributing to subacromial impingement syndrome.

Posterior capsular tightness is more common in overhead activities which increases the force on shoulder joint which may cause posterior capsular tightness along with rotator cuff tear. The active stabilizer for shoulder is rotator cuff which avoid the superior translation of humeral head during shoulder abduction due to weakness of rotator cuff along with posterior inferior capsular tightness the humeral head may translate superiorly and ultimately lead to SAIS in which rotator cuff tendon long head of biceps and subacromial bursa impinge between acromion superiorly and greater tubercle of humeral head inferiorly. Tears of the subscapularis tendon are mostly the result of a degenerative process, but less commonly, traumatic injury can result in acute subscapularis tearing. The most common mechanisms of subscapularis injury are hyperextension and external rotation of the shoulder.6 The infraspinatus (ISP) muscle, one of the rotator cuff muscles. Pain in the infraspinatus is most likely caused by repetitive motion involving the shoulder. Swimmers, tennis players, painters, and carpenters get it more frequently. It also becomes more likely as you get older.

The serratus anterior play an important role in prevention of shoulder impingement by lifting the acromion process in overhead activities. The most common pathologies of serratus anterior is serratus anterior dysfunction which may cause scapula winging.8 In GHIRD glenohumeral internal rotation deficit there is 18 to 20 degree of limitation along with glenohumeral horizontal adduction and incomplete humeral rotation can lead to posterior capsular tightness. Therefore, posterior capsular stretch is more effective intervention for posterior capsular tightness.AC joint is responsible for shoulder disability and pain in inactive patient and athletic activities including skiing, cycling and mostly in contact sports which contribute 9 percent approximately of AC joint damage with shoulder injuries. Impairment of AC joint effects range of motion, pain and weakness along with poor posture and these leads to restriction in overhead activities.

The most frequent causes are posterior capsular tightness and rotator cuff tear involve overhead movements such as swimming and volleyball and basketball, which have high-velocity pressures on the joint shoulder.

In non-operative management of subacromial impingement, anti-inflammatory mediction,subacromial injection of steriods, ultrasound, lifestyle changes, and physical therapy management is normally given. Physical therapy is used to reduce the pain and enhance the functioning of the SIS. Patients should attempt to discontinue overhead movements unless symptoms diminish.

A pragmatic posterior capsular stretch (PPCS) is designed to stretch the posterior capsule when it is in torsion.Pragmatic Posterior capsular stretch can effectively improve the functional movements and shoulder ROM of healthy young adults.16 Another popular stretch is the "sleeper stretch". There is a significant increase in posterior shoulder flexibility by sleeper stretch.Scapular movement is restricted while performing the sleeper stretch and accomplished by lying on the side to be stretched, elevating the humerus to 90° on the support surface, then passively internally rotating the shoulder with the opposite arm.

ELIGIBILITY:
Inclusion Criteria:

-Limitation in range of motion abduction or internal rotation or external rotation or reaching up behind the back or reaching behind down the neck are only one of the limitations in comparison with the unaffected joint.

A patient who fall in grade 1 and grade 2 of the shoulder mobility test of functional movement screening.

Exclusion Criteria:

-Patient with shoulder ligamentous instability Functional movement Screening score 0 or 3. Cancerous growth around the shoulder girdle Rheumatoid arthritis patients The patient has a recent fracture of less than the 6th-week duration or shoulder dislocation.

Long term use of steroids Cervical joint dysfunction, radicular pain. Systemic diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2021-12-24 (Estimated); Study Completion 2022-03-24 (Estimated)

PRIMARY OUTCOMES:
shoulder range of motion | 6 weeks
  shoulder range of motion will be measured in degrees by using digital inclinometer
shoulder pain | 6 weeks
  shoulder pain will be measured by numeric pain rating scale

SECONDARY OUTCOMES:
Shoulder related quality of life | 6 weeks
  quality of life will be measured by using HHIRS quality of life questionnaire
Shoulder disability | 6 weeks
  Shoulder disability will be measured by Shoulder Pain And Disability Index Urdu (SPADI-U)
satisfaction level of patient | 6 weeks
  satisfaction level of patient will be measured by Questionnaire for satisfaction level of patient receving this intervention

CONTACTS AND LOCATIONS:
Overall Officials: keramat ullah karamat, Ph.D.*, Principal Investigator — HHIRST
Locations (1):
- HHIRST, Mansehra, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
As per the decision of the research ethics committee.

REFERENCES:
- [Background] Michener LA, McClure PW, Karduna AR. Anatomical and biomechanical mechanisms of subacromial impingement syndrome. Clin Biomech (Bristol). 2003 Jun;18(5):369-79. doi: 10.1016/s0268-0033(03)00047-0. PMID 12763431
- [Background] Umer M, Qadir I, Azam M. Subacromial impingement syndrome. Orthop Rev (Pavia). 2012 May 9;4(2):e18. doi: 10.4081/or.2012.e18. Epub 2012 May 31. PMID 22802986
- [Background] Cools AM, Johansson FR, Borms D, Maenhout A. Prevention of shoulder injuries in overhead athletes: a science-based approach. Braz J Phys Ther. 2015 Sep-Oct;19(5):331-9. doi: 10.1590/bjpt-rbf.2014.0109. Epub 2015 Sep 1. PMID 26537804
- [Background] Lyons RP, Green A. Subscapularis tendon tears. J Am Acad Orthop Surg. 2005 Sep;13(5):353-63. doi: 10.5435/00124635-200509000-00009. PMID 16148361
- [Background] Johnson JE, Fullmer JA, Nielsen CM, Johnson JK, Moorman CT 3rd. Glenohumeral Internal Rotation Deficit and Injuries: A Systematic Review and Meta-analysis. Orthop J Sports Med. 2018 May 22;6(5):2325967118773322. doi: 10.1177/2325967118773322. eCollection 2018 May. PMID 29845083
- [Background] Keramat KU, Naveed Babur M. Pragmatic posterior capsular stretch and its effects on shoulder joint range of motion. BMJ Open Sport Exerc Med. 2020 Sep 9;6(1):e000805. doi: 10.1136/bmjsem-2020-000805. eCollection 2020. PMID 33062302
- [Background] Laudner KG, Sipes RC, Wilson JT. The acute effects of sleeper stretches on shoulder range of motion. J Athl Train. 2008 Jul-Aug;43(4):359-63. doi: 10.4085/1062-6050-43.4.359. PMID 18668168